CLINICAL TRIAL: NCT04425785
Title: Physical Exercise and Mental Wellbeing Rehabilitation for Acute Stress-induced Takotsubo Cardiomyopathy: The PLEASE Study
Acronym: PLEASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2-115-18
Record Dates: First submitted 2020-05-27; First posted 2020-06-11 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Takotsubo Cardiomyopathy
MeSH Terms: conditions — Takotsubo Cardiomyopathy | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomised controlled study. Takotsubo patients will be randomised into one of the following groups:
  Exercise Arm Cognitive Behavioural Arm Standard Clinical Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical Exercise Group (Experimental): A structured exercise program for 12 weeks
  Interventions: Other: Physical Exercise Program
- Cognitive Behavioural Therapy (Experimental): Cognitive Behavioural Therapy for 12 weeks
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Standard Clinical Care (No Intervention): Standard Clinical Care

INTERVENTIONS:
Other: Physical Exercise Program — A structured exercise program
  Arms: Physical Exercise Group
Behavioral: Cognitive Behavioural Therapy — A structured cognitive behavioural therapy program
  Arms: Cognitive Behavioural Therapy

SUMMARY:
Takotsubo cardiomyopathy presents like a heart attack and is typically triggered by intense emotional or physical stress. Recovery of this condition varies and many patients continue to suffer from symptoms such as fatigue and breathlessness for a protracted period after their event. Research conducted in our unit has found that the heart function does not recover fully as is commonly believed and that the energetic status of the heart remains impaired for an extended period of time. The purpose of our study is to establish whether following a structured exercise program or a mental wellbeing program compared to usual care for 12 weeks after an episode of Takotsubo will improve the energy status of the heart, their physical conditioning and improve the general mental wellbeing of patients.

DETAILED DESCRIPTION:
Acute takotsubo cardiomyopathy is characterised by sudden onset left ventricular dysfunction precipitated by major stress. The researchers have shown that recovery is more protracted than previously appreciated, and is associated with persistent major morbidity and a long-term heart failure phenotype. In the absence of any effective therapeutic options, the researchers propose a mechanistic three-arm pilot feasibility trial of early rehabilitation (standardised physical exercise training or cognitive behavioural therapy) versus current standard of care in patients who suffered a very recent episode of takotsubo cardiomyopathy. The primary end-point will be the restoration of cardiac energetic status assessed by 31P-magnetic resonance spectroscopy and the secondary end-points of cortisol awakening response, global longitudinal strain by echocardiography and the 6-minute walk test. If successful, this has the potential for rapid implementation into a large randomised clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* A patient who has recently suffered an episode of takotsubo cardiomyopathy within the last three weeks
* Participant who is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Any patient whose takotsubo cardiomyopathy was triggered by a physical illness that would preclude them for taking part in a physical exercise training program.
* Any patient who is not able or not willing to travel to the cardiovascular research facility for their study visits.
* Any patient who is not able to commit to a 12 week supervised training program.
* Inability to exercise on a cycle ergometer (i.e. use of walking aids or prosthetic limbs).
* Contraindication to magnetic resonance scanning such as an implantable cardiac device.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Cardiac Energetics | Within three weeks after diagnosis
  Cardiac Magnetic Resonance Imaging and Magnetic Resonance Spectroscopy
Cardiac Energetics | At completion of 12 weeks intervention
  Cardiac Magnetic Resonance Imaging and Magnetic Resonance Spectroscopy

SECONDARY OUTCOMES:
Left Ventricular Global Longitudinal Strain | Within three weeks after diagnosis
  Echocardiography
Left Ventricular Global Longitudinal Strain | At completion of 12 weeks intervention
  Echocardiography
Exercise Capacity | Within three weeks after diagnosis
  6 minute walk test and Cardiopulmonary Exercise Test
Exercise Capacity | At completion of 12 weeks intervention
  6 minute walk test and Cardiopulmonary Exercise Test
Mental status and Stress | Within three weeks after diagnosis
  Index of Mental Wellbeing and Cortisol Awakening Response
Mental status and Stress | At completion of 12 weeks intervention
  Index of Mental Wellbeing and Cortisol Awakening Response

CONTACTS AND LOCATIONS:
Overall Officials: Dana Dawson, MPhil, Principal Investigator — University of Aberdeen
Locations (1):
- Cardiac Research Facility, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prasad A, Lerman A, Rihal CS. Apical ballooning syndrome (Tako-Tsubo or stress cardiomyopathy): a mimic of acute myocardial infarction. Am Heart J. 2008 Mar;155(3):408-17. doi: 10.1016/j.ahj.2007.11.008. Epub 2008 Jan 31. PMID 18294473
- [Background] Templin C, Ghadri JR, Diekmann J, Napp LC, Bataiosu DR, Jaguszewski M, Cammann VL, Sarcon A, Geyer V, Neumann CA, Seifert B, Hellermann J, Schwyzer M, Eisenhardt K, Jenewein J, Franke J, Katus HA, Burgdorf C, Schunkert H, Moeller C, Thiele H, Bauersachs J, Tschope C, Schultheiss HP, Laney CA, Rajan L, Michels G, Pfister R, Ukena C, Bohm M, Erbel R, Cuneo A, Kuck KH, Jacobshagen C, Hasenfuss G, Karakas M, Koenig W, Rottbauer W, Said SM, Braun-Dullaeus RC, Cuculi F, Banning A, Fischer TA, Vasankari T, Airaksinen KE, Fijalkowski M, Rynkiewicz A, Pawlak M, Opolski G, Dworakowski R, MacCarthy P, Kaiser C, Osswald S, Galiuto L, Crea F, Dichtl W, Franz WM, Empen K, Felix SB, Delmas C, Lairez O, Erne P, Bax JJ, Ford I, Ruschitzka F, Prasad A, Luscher TF. Clinical Features and Outcomes of Takotsubo (Stress) Cardiomyopathy. N Engl J Med. 2015 Sep 3;373(10):929-38. doi: 10.1056/NEJMoa1406761. PMID 26332547
- [Background] Tornvall P, Collste O, Ehrenborg E, Jarnbert-Petterson H. A Case-Control Study of Risk Markers and Mortality in Takotsubo Stress Cardiomyopathy. J Am Coll Cardiol. 2016 Apr 26;67(16):1931-6. doi: 10.1016/j.jacc.2016.02.029. PMID 27102508
- [Background] Stiermaier T, Moeller C, Oehler K, Desch S, Graf T, Eitel C, Vonthein R, Schuler G, Thiele H, Eitel I. Long-term excess mortality in takotsubo cardiomyopathy: predictors, causes and clinical consequences. Eur J Heart Fail. 2016 Jun;18(6):650-6. doi: 10.1002/ejhf.494. Epub 2016 Mar 14. PMID 26990821
- [Background] Scally C, Rudd A, Mezincescu A, Wilson H, Srivanasan J, Horgan G, Broadhurst P, Newby DE, Henning A, Dawson DK. Persistent Long-Term Structural, Functional, and Metabolic Changes After Stress-Induced (Takotsubo) Cardiomyopathy. Circulation. 2018 Mar 6;137(10):1039-1048. doi: 10.1161/CIRCULATIONAHA.117.031841. Epub 2017 Nov 11. PMID 29128863
- [Background] Isogai T, Matsui H, Tanaka H, Fushimi K, Yasunaga H. Early beta-blocker use and in-hospital mortality in patients with Takotsubo cardiomyopathy. Heart. 2016 Jul 1;102(13):1029-35. doi: 10.1136/heartjnl-2015-308712. Epub 2016 Feb 15. PMID 26879240
- [Background] Singh K, Carson K, Usmani Z, Sawhney G, Shah R, Horowitz J. Systematic review and meta-analysis of incidence and correlates of recurrence of takotsubo cardiomyopathy. Int J Cardiol. 2014 Jul 1;174(3):696-701. doi: 10.1016/j.ijcard.2014.04.221. Epub 2014 Apr 26. PMID 24809923
- [Background] Kitzman DW, Brubaker PH, Herrington DM, Morgan TM, Stewart KP, Hundley WG, Abdelhamed A, Haykowsky MJ. Effect of endurance exercise training on endothelial function and arterial stiffness in older patients with heart failure and preserved ejection fraction: a randomized, controlled, single-blind trial. J Am Coll Cardiol. 2013 Aug 13;62(7):584-92. doi: 10.1016/j.jacc.2013.04.033. Epub 2013 May 9. PMID 23665370
- [Background] Coats AJ, Adamopoulos S, Radaelli A, McCance A, Meyer TE, Bernardi L, Solda PL, Davey P, Ormerod O, Forfar C, et al. Controlled trial of physical training in chronic heart failure. Exercise performance, hemodynamics, ventilation, and autonomic function. Circulation. 1992 Jun;85(6):2119-31. doi: 10.1161/01.cir.85.6.2119. PMID 1591831
- [Background] O'Connor CM, Whellan DJ, Lee KL, Keteyian SJ, Cooper LS, Ellis SJ, Leifer ES, Kraus WE, Kitzman DW, Blumenthal JA, Rendall DS, Miller NH, Fleg JL, Schulman KA, McKelvie RS, Zannad F, Pina IL; HF-ACTION Investigators. Efficacy and safety of exercise training in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1439-50. doi: 10.1001/jama.2009.454. PMID 19351941
- [Background] Hegde SM, Claggett B, Shah AM, Lewis EF, Anand I, Shah SJ, Sweitzer NK, Fang JC, Pitt B, Pfeffer MA, Solomon SD. Physical Activity and Prognosis in the TOPCAT Trial (Treatment of Preserved Cardiac Function Heart Failure With an Aldosterone Antagonist). Circulation. 2017 Sep 12;136(11):982-992. doi: 10.1161/CIRCULATIONAHA.117.028002. Epub 2017 Jun 21. PMID 28637881
- [Background] Pandey A, Garg S, Khunger M, Darden D, Ayers C, Kumbhani DJ, Mayo HG, de Lemos JA, Berry JD. Dose-Response Relationship Between Physical Activity and Risk of Heart Failure: A Meta-Analysis. Circulation. 2015 Nov 10;132(19):1786-94. doi: 10.1161/CIRCULATIONAHA.115.015853. Epub 2015 Oct 5. PMID 26438781
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Smolderen KG, Buchanan DM, Gosch K, Whooley M, Chan PS, Vaccarino V, Parashar S, Shah AJ, Ho PM, Spertus JA. Depression Treatment and 1-Year Mortality After Acute Myocardial Infarction: Insights From the TRIUMPH Registry (Translational Research Investigating Underlying Disparities in Acute Myocardial Infarction Patients' Health Status). Circulation. 2017 May 2;135(18):1681-1689. doi: 10.1161/CIRCULATIONAHA.116.025140. Epub 2017 Feb 16. PMID 28209727
- [Background] Rozanski A, Blumenthal JA, Davidson KW, Saab PG, Kubzansky L. The epidemiology, pathophysiology, and management of psychosocial risk factors in cardiac practice: the emerging field of behavioral cardiology. J Am Coll Cardiol. 2005 Mar 1;45(5):637-51. doi: 10.1016/j.jacc.2004.12.005. PMID 15734605
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Background] Rosengren A, Hawken S, Ounpuu S, Sliwa K, Zubaid M, Almahmeed WA, Blackett KN, Sitthi-amorn C, Sato H, Yusuf S; INTERHEART investigators. Association of psychosocial risk factors with risk of acute myocardial infarction in 11119 cases and 13648 controls from 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):953-62. doi: 10.1016/S0140-6736(04)17019-0. PMID 15364186
- [Background] Blumenthal JA, Sherwood A, Babyak MA, Watkins LL, Waugh R, Georgiades A, Bacon SL, Hayano J, Coleman RE, Hinderliter A. Effects of exercise and stress management training on markers of cardiovascular risk in patients with ischemic heart disease: a randomized controlled trial. JAMA. 2005 Apr 6;293(13):1626-34. doi: 10.1001/jama.293.13.1626. PMID 15811982
- [Background] Chen X, Lee G, Maher BS, Fanous AH, Chen J, Zhao Z, Guo A, van den Oord E, Sullivan PF, Shi J, Levinson DF, Gejman PV, Sanders A, Duan J, Owen MJ, Craddock NJ, O'Donovan MC, Blackman J, Lewis D, Kirov GK, Qin W, Schwab S, Wildenauer D, Chowdari K, Nimgaonkar V, Straub RE, Weinberger DR, O'Neill FA, Walsh D, Bronstein M, Darvasi A, Lencz T, Malhotra AK, Rujescu D, Giegling I, Werge T, Hansen T, Ingason A, Noethen MM, Rietschel M, Cichon S, Djurovic S, Andreassen OA, Cantor RM, Ophoff R, Corvin A, Morris DW, Gill M, Pato CN, Pato MT, Macedo A, Gurling HM, McQuillin A, Pimm J, Hultman C, Lichtenstein P, Sklar P, Purcell SM, Scolnick E, St Clair D, Blackwood DH, Kendler KS; GROUP investigators; International Schizophrenia Consortium. GWA study data mining and independent replication identify cardiomyopathy-associated 5 (CMYA5) as a risk gene for schizophrenia. Mol Psychiatry. 2011 Nov;16(11):1117-29. doi: 10.1038/mp.2010.96. Epub 2010 Sep 14. PMID 20838396
- [Background] Ashbrook DG, Williams RW, Lu L, Hager R. A cross-species genetic analysis identifies candidate genes for mouse anxiety and human bipolar disorder. Front Behav Neurosci. 2015 Jul 1;9:171. doi: 10.3389/fnbeh.2015.00171. eCollection 2015. PMID 26190982
- [Background] McCalmon SA, Desjardins DM, Ahmad S, Davidoff KS, Snyder CM, Sato K, Ohashi K, Kielbasa OM, Mathew M, Ewen EP, Walsh K, Gavras H, Naya FJ. Modulation of angiotensin II-mediated cardiac remodeling by the MEF2A target gene Xirp2. Circ Res. 2010 Mar 19;106(5):952-60. doi: 10.1161/CIRCRESAHA.109.209007. Epub 2010 Jan 21. PMID 20093629
- [Background] Pison L, De Vusser P, Mullens W. Apical ballooning in relatives. Heart. 2004 Dec;90(12):e67. doi: 10.1136/hrt.2004.046813. PMID 15547001
- [Background] Kumar G, Holmes DR Jr, Prasad A. "Familial" apical ballooning syndrome (Takotsubo cardiomyopathy). Int J Cardiol. 2010 Oct 29;144(3):444-5. doi: 10.1016/j.ijcard.2009.03.078. Epub 2009 Apr 17. PMID 19375184
- [Background] Sharkey SW, Lips DL, Pink VR, Maron BJ. Daughter-mother tako-tsubo cardiomyopathy. Am J Cardiol. 2013 Jul 1;112(1):137-8. doi: 10.1016/j.amjcard.2013.02.063. Epub 2013 Apr 2. PMID 23561588
- [Background] Caretta G, Robba D, Vizzardi E, Bonadei I, Raddino R, Metra M. Tako-tsubo cardiomyopathy in two sisters: a chance finding or familial predisposition? Clin Res Cardiol. 2015 Jul;104(7):614-6. doi: 10.1007/s00392-015-0837-0. Epub 2015 Mar 6. No abstract available. PMID 25743177
- [Background] Lyon AR, Bossone E, Schneider B, Sechtem U, Citro R, Underwood SR, Sheppard MN, Figtree GA, Parodi G, Akashi YJ, Ruschitzka F, Filippatos G, Mebazaa A, Omerovic E. Current state of knowledge on Takotsubo syndrome: a Position Statement from the Taskforce on Takotsubo Syndrome of the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2016 Jan;18(1):8-27. doi: 10.1002/ejhf.424. Epub 2015 Nov 9. PMID 26548803
- [Background] Madhavan M, Prasad A. Proposed Mayo Clinic criteria for the diagnosis of Tako-Tsubo cardiomyopathy and long-term prognosis. Herz. 2010 Jun;35(4):240-3. doi: 10.1007/s00059-010-3339-x. PMID 20582391
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Barwell ND, Malkova D, Moran CN, Cleland SJ, Packard CJ, Zammit VA, Gill JM. Exercise training has greater effects on insulin sensitivity in daughters of patients with type 2 diabetes than in women with no family history of diabetes. Diabetologia. 2008 Oct;51(10):1912-9. doi: 10.1007/s00125-008-1097-6. Epub 2008 Jul 29. PMID 18663427
- [Background] Ridgway N, Williams C. Cognitive behavioural therapy self-help for depression: an overview. J Ment Health. 2011 Dec;20(6):593-603. doi: 10.3109/09638237.2011.613956. PMID 22126636
- [Background] Williams C, McClay CA, Matthews L, McConnachie A, Haig C, Walker A, Morrison J. Community-based group guided self-help intervention for low mood and stress: randomised controlled trial. Br J Psychiatry. 2018 Feb;212(2):88-95. doi: 10.1192/bjp.2017.18. PMID 29436324
- [Background] Dawson DK, Neil CJ, Henning A, Cameron D, Jagpal B, Bruce M, Horowitz J, Frenneaux MP. Tako-Tsubo Cardiomyopathy: A Heart Stressed Out of Energy? JACC Cardiovasc Imaging. 2015 Aug;8(8):985-7. doi: 10.1016/j.jcmg.2014.10.004. Epub 2014 Nov 1. No abstract available. PMID 25499134
- [Background] Scally C, Ahearn T, Rudd A, Neil CJ, Srivanasan J, Jagpal B, Horowitz J, Frenneaux M, Dawson DK. Right Ventricular Involvement and Recovery After Acute Stress-Induced (Tako-tsubo) Cardiomyopathy. Am J Cardiol. 2016 Mar 1;117(5):775-80. doi: 10.1016/j.amjcard.2015.11.057. Epub 2015 Dec 13. PMID 26782339
- [Background] Schwarz K, Ahearn T, Srinivasan J, Neil CJ, Scally C, Rudd A, Jagpal B, Frenneaux MP, Pislaru C, Horowitz JD, Dawson DK. Alterations in Cardiac Deformation, Timing of Contraction and Relaxation, and Early Myocardial Fibrosis Accompany the Apparent Recovery of Acute Stress-Induced (Takotsubo) Cardiomyopathy: An End to the Concept of Transience. J Am Soc Echocardiogr. 2017 Aug;30(8):745-755. doi: 10.1016/j.echo.2017.03.016. Epub 2017 Jun 7. PMID 28599831
- [Derived] Gamble DT, Ross J, Khan H, Cheyne L, Rudd A, Srivanasan J, Horgan G, Hogg D, Myint PK, Newby DE, Williams C, Gray SR, Dawson D. Physical Exercise or Cognitive Behavioral Therapy for Takotsubo Cardiomyopathy: A Randomized Controlled Trial. Circ Heart Fail. 2025 Dec 3:e013229. doi: 10.1161/CIRCHEARTFAILURE.125.013229. Online ahead of print. PMID 41332388